CLINICAL TRIAL: NCT02776826
Title: World Bleeding Disorders Registry Pilot Phase
Brief Title: World Bleeding Disorders Registry Pilot Study
Acronym: WBDR
Status: Completed | Type: Observational
Sponsor: World Federation of Hemophilia (Other)
Responsible Party: Sponsor
Other Study IDs: WBDR Pilot Phase
Record Dates: First submitted 2016-05-11; First posted 2016-05-18 (Estimated); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Hemophilia A and B
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Months
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The World Federation of Hemophilia (WFH) is conducting the pilot phase of an international, observational, World Bleeding Disorders Registry (WBDR). This pilot phase will assess the feasibility of conducting an expanded WBDR to more centres with a more comprehensive case report form, around the world.

DETAILED DESCRIPTION:
The pilot phase of the WBDR is an observational disease registry of patients with hemophilia. Forty hemophilia treatment centres (HTCs), of varying levels of economic development (emerging, mid-level and established), that have data entry capabilities and the ability to obtain the required data on patients in English, were invited to participate in the pilot phase. Participating HTCs will complete a Minimal Data Set (MDS) of data on approximately 10 patients each.

A series of performance indicators have been identified by the Steering committee and will be used to assess the feasibility of expanding the pilot phase to the WBDR. The performance indicators include: proportion of HTCs invited that are willing to participate; proportion of participating HTCs who successfully obtain necessary regulatory approvals; proportion of patients approached who consent to participate; proportion of enrolled patients on which data collection and database entry is successful.

ELIGIBILITY:
Inclusion Criteria:

* Patients of participating Hemophilia Treatment Centres with Hemophilia A or B.
* Ability to provide data in English

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Hemophilia A or B, who are patients of participating Hemophilia Treatment Centres.
Sampling Method: Non-Probability Sample
Enrollment: 356 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Proportion of HTCs which agree to participate in the pilot phase of the WBDR | 6 months
  This is be measured by the number of HTCs who agree to participate, divided by the number of HTCs invited.
Proportion of participating HTCs who successfully obtain necessary regulatory approval | 6 months
  This will be measured by the number of HTCs who obtain approval, divided by the number of HTCs who have agreed to participate in the pilot phase of the WBDR.
Proportion of patients who agree to participate in this pilot phase of the WBDR. | 6 months
  This will be measured by the number of patients who provided consent to participate, divided by the number of patients who were approached to participate.
Proportion of enrolled patients on which data collection and database entry is successful. | 6 months
  This will be measured by the number of patients on who data is collected and entered successfully into the database, divided by the number of patients who are enrolled in the pilot phase of the WBDR.